CLINICAL TRIAL: NCT03369405
Title: Thyroid Insufficiency as a Modifying Factor for Chronic Periodontitis
Brief Title: Thyroid Disease and Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Dr. Lisa Yerke, Clinical Associate Professor, Department of Periodontics and Endodontics, University at Buffalo
Other Study IDs: STUDY00001811
Record Dates: First submitted 2017-11-28; First posted 2017-12-12 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Diseases; Chronic Periodontitis
Keywords: periodontitis; hypothyroidism
MeSH Terms: conditions — Thyroid Diseases; Chronic Periodontitis; Periodontitis; Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontally healthy patients: Patients that have no history of periodontal treatment and that have been scheduled for routine prophylaxis appointments in the predoctoral clinics at the School of Dental Medicine, University at Buffalo.
  Interventions: Other: NO intervention, patient records review only
- Periodontitis, group 1: Patients that have been referred from the pre-doctoral dental clinics to the Postgraduate Periodontics clinic for advanced periodontal disease. Clinical attachment loss, pain, mobility, bleeding, suppuration, and probing depths > 4 mm more likely to be prevalent.
  Interventions: Other: NO intervention, patient records review only
- Periodontitis, group 2: Patients referred to a faculty practice periodontist over the course of his clinical career due to chronic periodontitis that could not be treated by the referring general dentist. Clinical attachment loss, pain, mobility, bleeding, suppuration, and probing depths > 4 mm more likely to be prevalent.
  Interventions: Other: NO intervention, patient records review only

INTERVENTIONS:
Other: NO intervention, patient records review only — There is no intervention - the three study groups are created by utilizing three unique sets of search criteria for the patient records review.

SUMMARY:
Currently, the investigators are unaware of any previous studies that have analyzed the relationship between the prevalence of thyroid disease and chronic periodontitis among adults utilizing a retrospective, cross-sectional design. This study will review approximately 2000 patient records and compare the prevalence of thyroid disease in three groups with increasing severity of chronic periodontitis.

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional patient records review study. Only records with subjects that were 35 years or older and have been active patients of the School of Dental Medicine, University at Buffalo will be included. Three individual searches with three distinct patient criteria will be conducted to obtain records from subjects in three populations with different degrees of periodontal disease. All subjects that qualify the eligibility criteria will be selected. The IT Department has access to select the subjects according to the eligibility criteria without requiring access to the physical patient record. The three subject groups are:

1. Periodontally healthy patients: Patients with a D1110 or D1111 (adult prophylaxis including those with 6 or fewer teeth) treatment code, seen by a 3rd or 4th year pre-doctoral dental student. Excludes all charts that have ever had a U4990 (Perio case) treatment code. Patient is 35 years or older relative to 1/1/2016.
2. Patients with a history of advanced periodontal treatment, group 1: All patients treated in the Postgraduate Periodontics department by a periodontics resident between 1/1/2000 - 12/31/2017. Patients presenting for treatment of chronic periodontitis will be included while those patients presenting to the clinic for other reasons, such as crown lengthening procedures, will be labeled as such. All patients selected will be 35 years or older at time of initial exam.
3. Patients with history of advanced periodontal treatment, group 2: All patients ever treated in the private faculty practice of one periodontist, that were still active patients during between 1/1/16 - 12/31/16. Only those 35 years and older were included. Patients presenting for treatment of chronic periodontitis will be included while those patients presenting to the clinic for other reasons, such as crown lengthening procedures, will be labeled as such.

All duplicates within a group will be excluded (e.g. patients may have had a D1110 code more than once per year). These 3 subject search criteria should yield a sufficient number of patient records for statistical analysis.

All patient records will be reviewed and data will be collected and recorded in an electronic Microsoft Excel database file that is saved on an encrypted flash drive. The only patient identifier recorded will be the patient records number. Once data collection is complete, or at a maximum of 3 years from the start of the study, all identifying information will be deleted and only de-identified data saved on a separate electronic file will be analyzed. No code key will be required.

Data will be analyzed using ANOVA (F-test). If multiple variables are used, analysis will be by using generalized estimating equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

* Active patient of the School of Dental Medicine, University at Buffalo.
* The remaining eligibility criteria varies between the three distinct subject populations, which are noted below. All eligibility criteria is selected for by an electronic search of patient records performed by the IT Department at the School of Dental Medicine, University at Buffalo.

  1. Periodontally healthy patients:

     1. A treatment code of D1110 or D111 was processed at least once but excluding patients that were ever assigned a treatment code of U4990
     2. A 3rd or 4th year pre-doctoral dental student provider
     3. 35 years or older as of 1/1/2016
     4. Patient presented to clinic between 1/1/2016-12/31/2016
  2. Patients with history of advanced periodontal treatment, group 1:

     1. All patients presenting to the Postgraduate Periodontics Department at UB and being seen by a periodontics resident
     2. Time period between 1/1/2000-12/31/2017
     3. Patients will be 35 years or older at time of initial exam
     4. Patients presenting for reasons other than chronic periodontitis treatment (e.g. crown lengthening) will be labeled as such.
  3. Patients with history of advanced periodontal treatment, group 2:

     1. All patients treated in the faculty practice of one periodontist that remained active patients during the time period 1/1/2016-12/31-2016
     2. All patients were 35 years or older at time of initial exam

Duplicates within groups are eliminated.

Exclusion Criteria:

* inadequate data from records

Note: the majority of patient records selected by the search criteria done electronically by the IT department will be included in the study, since the search criteria very closely overlaps the overall study criteria

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is sampled from the patient records available at the School of Dental Medicine, University at Buffalo, State University of New York. The patient records reviewed will be of patients seen in the predoctoral as well as postgraduate clinics.
  The third group population is sampled from the patient records available from the faculty practice of one provider located at the University of Buffalo, State University of New York
Sampling Method: Non-Probability Sample
Enrollment: 4965 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Thyroid disease prevalence | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  The presence or absence of thyroid medication in the patient record will be used as a surrogate marker for thyroid disease presence or absence.

SECONDARY OUTCOMES:
smoking history | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  Smoking history will be determined from the Medical Questionnaire form in the patient records.
diabetes disease prevalence | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  The Medical Questionnaire and the Medication List in the patient records will be referenced to determine the presence of diabetes.
Periodontal Probing Depths 5mm or greater | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  Number of teeth that have one or more sites that contain a 5mm or greater pocket, recorded in periodontal chart
Periodontal Probing Depths 6mm or greater | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  Number of teeth that have one or more sites that contain a 6mm or greater pocket, recorded in periodontal chart
Teeth | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  Total number of teeth, recorded in periodontal chart
proton pump inhibitor use | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  The Medication List in the patient records will be referenced to determine any history of proton pump inhibitor use.
Plaque Score | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  Percentage of tooth surfaces positive for plaque out of total tooth surfaces
Hormone replacement therapy | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  The presence or absence of hormone supplementation (birth control or hormone replacement therapy included)
bisphosphonate use | Assessed at one time point only, during patient's initial exam noted in patient records (cross-sectional study).
  The Medication List in the patient records will be referenced to determine any history of bisphosphonate use.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No